CLINICAL TRIAL: NCT01929395
Title: A Study to Evaluate the Use of Supine MRI Images in Breast Conserving Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Richard J. Barth,Jr., Section Chief, General Surgery, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: D0928; NCI-2011-03481 (Other: NCI)
Record Dates: First submitted 2013-04-05; First posted 2013-08-27 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Conserving Surgery; Breast diagnostics; Breast imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 addition of supine MRI to conventional imaging (Active Comparator): Arm 1 objective will be to determine whether the addition of supine MRI to conventional imaging with mammography and or sonography and prone MRI will result in a lower positive margin rate in patients undergoing breast conserving surgery.
  Interventions: Device: Supine MRI
- Arm 2 randomize to SOC vs supine MRI + SOC (Active Comparator): Arm 2 of the study patients with non-palpable invasive breast cancer or DCIS who desire breast conservation will be randomized to either a usual care group, or a group receiving a supine MRI in addition to conventional imaging (mammogram and prone MRI) and undergoing breast cancer resection without the wire localization technique.
  Interventions: Device: Supine MRI

INTERVENTIONS:
Device: Supine MRI — A limitation of MRI studies of the breast is that MRI exams are performed with the patient prone and the breasts in a pendant position, which is markedly different than the position of the breast when the patient is supine on the Operating Room table. The spatial information the surgeon receives from the prone MRI about the site of the tumor in the breast is hard to mentally translate into the actual site of the tumor in the breast of a supine patient prepared for surgery.

SUMMARY:
This is a 2 Phase study. In the first phase of the study, patients with palpable invasive breast cancer underwent pre-operative supine MRI and optical scanning in the surgical position. In the second phase of the study, patients with non-palpable invasive breast cancer or DCIS who desire breast conservation will be randomized to either a usual care group, or a group receiving a supine MRI in addition to conventional imaging (mammogram and prone MRI) and undergoing breast cancer resection without the wire localization technique.

DETAILED DESCRIPTION:
We propose to use a novel technique (optical scanning) to correlate the supine MRI image to the surgical position in the OR and then to confirm and extend the Japanese study described above. In the first phase of the study, 5-25 patients with palpable invasive breast cancer will undergo pre-operative supine MRI and optical scanning in the surgical position. The purpose of this phase will be ensure that the images created from the optical scanner-adjusted supine MRI images closely correspond to the location of the palpable tumors in these breasts. All patients will then have their tumor resected using the standard method of either palpation or image guided wire localization. The first phase has been completed.

In the second phase of the study, patients with non-palpable invasive breast cancer or DCIS who desire breast conservation will be randomized to either a usual care group, or a group receiving a supine MRI in addition to conventional imaging (mammogram and prone MRI) and undergoing breast cancer resection without the wire localization technique.

Our secondary objectives will be to determine:

1. whether there are differences between the two groups in the volume of breast tissue removed.
2. whether diagnostic information obtained from a supine MRI is equivalent to that obtained from the prone MRI.

ELIGIBILITY:
Inclusion Criteria Phase 1

1. Age greater than/equal to 18 years
2. Histologic diagnosis of palpable invasive breast cancer or ductal carcinoma in situ
3. Patient desire to undergo breast surgery

3. Patients will have provided informed consent to participate, documented by their signature on the study consent form 4. The cancer enhances on breast MRI imaging.

Inclusion Criteria Phase 2

1. Age greater than/equal to 18 years
2. Histologic diagnosis of invasive breast cancer or ductal carcinoma in situ
3. The tumor is visible and enhances on prone MRI and is >1 cm in greatest diameter.
4. . Determination by the surgeon that the neoplasm is non-palpable.A patient with a palpable hematoma from core biopsy, but a non-palpable neoplasm, will be eligible for study
5. Patient desire to undergo breast conserving surgery
6. Patients will have provided informed consent to participate, documented by their signature on the study consent form.The process of informed consent will be documented in the medical record and a copy of the signed consent form will be given to the patient.

Exclusion Criteria (Phases 1 and 2)

1. Absolute contraindication to MRI, including presence of implanted electrical device (pacemaker or neurostimulator), aneurysm clip or metallic foreign body in or near eyes
2. Severe claustrophobia
3. Contraindication to use of gadolinium based intravenous contrast, including life threatening allergy or compromised renal function (creatinine > 2.0)
4. History of median sternotomy
5. Pregnancy (Patient attestation that they are not pregnant will be acceptable, as per standard, as per standard policy for MRIs at DHMC).
6. Multicentric breast cancer, defined as two or more tumors in different quadrants of the breast. An eligibility worksheet will be completed for each patient prior to enrollment and will be signed and dated by the surgeon investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants from Phase 1 participated in Phase 2
Groups:
- Phase 1: Addition of Supine MRI to Conventional Imaging; Phase 2: Addition of Supine MRI to Conventional Imaging: Pre-operative supine MRI with intraoperative optical scanning and tracking (group MRI)
- Phase 2: Conventional Imaging (SOC): Wire localized (group WL) partial mastectomy
Period: Overall Study
Arm/Group | Phase 1: Addition of Supine MRI to Conventional Imaging | Phase 2: Addition of Supine MRI to Conventional Imaging | Phase 2: Conventional Imaging (SOC)
Started | 19 | 70 | 70
Completed | 18 | 69 | 69
Not Completed | 1 | 1 | 1
Not completed — Did not complete - non-related toxicity | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Screen Fail | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Addition of Supine MRI to Conventional Imaging | Phase 2: Addition of Supine MRI to Conventional Imaging | Phase 2: Conventional Imaging (SOC) | Total
Number analyzed (Participants) | 18 | 69 | 69 | 156
Age, Customized [Count of Participants; unit: Participants]
  >=18 years | 18 | 69 | 69 | 156
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 69 | 69 | 156
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 18 | 69 | 69 | 156
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 69 | 69 | 156

OUTCOME MEASURES:

1. Primary Outcome: The Mean Distance Between the Image-defined and Palpation-defined Edges of the Tumor.
Description: Mean calculated from differences in precise distances from the nipple to the superior, inferior, medial and lateral edges of the tumor as determined from the adjusted MRI images and conventional MRI.
Time Frame: From baseline MRI to intraoperative measurements: 30 days
Measure: Mean (Full Range); unit: mm
Arm/Group | Phase 1: Addition of Supine MRI to Conventional Imaging
Number analyzed (Participants) | 18
mm | 7.2 [0 to 19]

2. Primary Outcome: To Determine Whether the Addition of Supine MRI to Conventional Imaging With Mammography and Prone MRI Results in a Lower Positive Margin Rate in Patients Undergoing Breast-conserving Surgery.
Description: The primary analysis consists of computing the positive margin rate observed in the two groups and comparing them with a chi-squared test and finally comparing the proportion of patients with positive margins in the two groups based on study criteria.
Time Frame: 30 days from surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Addition of Supine MRI to Conventional Imaging | Phase 2: Conventional Imaging (SOC)
Number analyzed (Participants) | 68 | 69
Participants | 8 | 16

3. Secondary Outcome: Differences Between the Two Groups in the Volume of Breast Tissue Removed
Description: The mean specimen volumes to be compared using t - statistics. The concordance between lesion volumes identified on the supine MRI images and the prone MRI images will be evaluated through correlation and regression analysis.
Time Frame: 30 days from surgery
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Phase 2: Addition of Supine MRI to Conventional Imaging | Phase 2: Conventional Imaging (SOC)
Number analyzed (Participants) | 68 | 69
ml | 74 (33.9) | 69.8 (25.1)

ADVERSE EVENTS:
Time Frame: From the inception of Phase 1 (baseline) to end of intervention for Phase 2: 7 years
Description: Regular investigator assessment and regular laboratory testing
Arm/Group | Phase 1: Addition of Supine MRI to Conventional Imaging | Phase 2: Addition of Supine MRI to Conventional Imaging | Phase 2: Conventional Imaging (SOC)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/69 | 1/69
Other Adverse Events (participants affected / at risk) | 0/18 | 0/69 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Addition of Supine MRI to Conventional Imaging (N=18) | Phase 2: Addition of Supine MRI to Conventional Imaging (N=69) | Phase 2: Conventional Imaging (SOC) (N=69)
Hematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) — Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT01929395/Prot_SAP_000.pdf